CLINICAL TRIAL: NCT00031772
Title: Enhancing Well-Being During Breast Cancer Recurrence. SWOG Study S9832.
Brief Title: S9832: Effectiveness of Telephone Counseling By Breast Cancer Survivors on the Well-Being of Women With Recurrent Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CDR0000069225; S9832 (Other: SWOG); NCI-P02-0209 (Other: NCI); U10CA037429 (NIH)
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Breast Cancer; Psychosocial Effects of Cancer and Its Treatment
Keywords: recurrent breast cancer; psychosocial effects of cancer and its treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Standard level of support after recurrence diagnosis
- Intervention (Experimental): Phone intervention for patients experiencing first recurrence with quality of life questionnaires, psychosocial assessment and care.
  Interventions: Procedure: psychosocial assessment and care

INTERVENTIONS:
Procedure: psychosocial assessment and care — Questionnaire and telephone intervention
  Arms: Intervention

SUMMARY:
RATIONALE: Telephone counseling by breast cancer survivors may enhance the well-being and quality of life of women who have recurrent breast cancer.

PURPOSE: Randomized clinical trial to study the effectiveness of telephone counseling by breast cancer survivors on the well-being of women who have recurrent breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether telephone counseling delivered by breast cancer survivors enhances the well-being of women with recurrent breast cancer.
* Determine the impact of sociodemographic, clinical, and psychosocial predictors of well-being in these patients.
* Determine the changes in well-being over time since disease recurrence in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to age (under 50 vs 50 and over), time since initial diagnosis (less than 2 years vs 2 years or more), and recurrence site (soft tissue without bone vs soft tissue with bone vs visceral). Patients are randomized to one of two study arms.

* Arm I (control arm): Patients receive the standard level of support by continuing to use existing resources. Patients receive written materials from the counseling group at 6 months.
* Arm II (intervention arm): Patients receive weekly telephone counseling sessions by breast cancer survivors over 4 weeks for a total of 4-8 sessions. Patients receive written materials from the counseling group after the first session.

In both arms, quality of life is assessed at baseline and at 3 and 6 months.

PROJECTED ACCRUAL: A total of 300 patients (150 per study arm) will be accrued for this study within 30 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Received prior definitive surgical treatment for stage I-IIIa breast cancer with or without adjuvant chemotherapy, hormonal therapy, and/or radiotherapy
* No more than 56 days since diagnosis of first recurrence

  * Any distant metastatic site, chest wall recurrence, scar recurrence, or nodal recurrence
  * No ipsilateral breast tumor recurrence after lumpectomy or isolated contralateral new primary breast tumors
* Receiving or planning to receive first therapy for recurrence

  * No prior therapy for this recurrence except surgical treatment for in-breast relapse after lumpectomy or local palliative radiotherapy
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* Not specified

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No psychiatric diagnosis that would preclude study
* Must be able to read and understand English

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* See Disease Characteristics

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 1998-07; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Assess effectiveness of a telephone intervention delivered by breast cancer survivors on well-being of patients experiencing a first recurrence of breast cancer | 6 months

SECONDARY OUTCOMES:
Examine impact of sociodemographic, clinical, and psychosocial predictors of well-being in patients experiencing a first recurrence of breast cancer. | 6 months
Examine changes in well-being over time since recurrence | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Gotay, PhD, Study Chair — University of Hawaii Cancer Research Center
Locations (108):
- United States (107):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Carl T. Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Veterans Affairs Medical Center - West Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Van Nuys Breast Center, Van Nuys, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - MBCCOP-Howard University Cancer Center, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Western New York Urology Associates, Buffalo, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - OHSU Cancer Institute, Portland, Oregon
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - Eastern Virginia Medical School, Norfolk, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
- British Columbia Cancer Agency, Vancouver, British Columbia, Canada

REFERENCES:
- [Result] Gotay CC, Moinpour CM, Unger JM, Jiang CS, Coleman D, Martino S, Parker BJ, Bearden JD, Dakhil S, Gross HM, Lippman S, Albain KS. Impact of a peer-delivered telephone intervention for women experiencing a breast cancer recurrence. J Clin Oncol. 2007 May 20;25(15):2093-9. doi: 10.1200/JCO.2006.07.4674. PMID 17513815
- [Result] Gotay CC, Moinpour CM, Jiang CS, et al.: Enhancing well-being during breast cancer recurrence: preliminary findings from a phase III study. [Abstract] Breast Cancer Res Treat 88 (Suppl 1): A-3080, 2004.